CLINICAL TRIAL: NCT01226329
Title: The Right Question Project-Mental Health: An Intervention to Increase Engagement and Retention in Mental Health Care
Acronym: RQP-MH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Margarita Alegria, PhD, Chief, Disparities Research Unit, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CHA-IRB00329/07/08; P60MD002261-03 (NIH)
Record Dates: First submitted 2010-09-16; First posted 2010-10-22 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Mental Disorders
Keywords: Minority Groups; Decision Making; Patient Participation; Mental Health Services; retention; attendance; patient activation; Hispanic Americans; patient-provider communication
MeSH Terms: conditions — Mental Disorders; Patient Participation | interventions — Self-Management; Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RQP-MH (Experimental): Participants in the intervention arm will receive three Patient Activation and Self-Management education sessions, plus a fourth booster session if they show difficulty mastering the content of the first three trainings.
  Interventions: Behavioral: Right Question Project - Mental Health (RQP-MH)
- Comparison Group (Active Comparator): Participants in this arm will receive a pamphlet in either Spanish or English called "Managing Your Mental Health Care."
  Interventions: Behavioral: Pamphlet

INTERVENTIONS:
Behavioral: Right Question Project - Mental Health (RQP-MH) — The RQP-MH trainings each take approximately 45 minutes to complete and are delivered approximately three weeks apart. The manualized intervention uses a Question Formulation Technique (QFT) and a Framework for Active Decision-Making (FADM). The QFT consists of asking patients to generate and revise questions to obtain more informative answers from their providers. The FADM teaches participants to identify questions that will help them consider their role in a decision, the process of decision-making, and the reasons behind a decision. All intervention sessions will be taught by a bachelors-level "Care Manager."
  Other Names: Patient Activation and Self-Management (PASM) intervention
  Arms: RQP-MH
Behavioral: Pamphlet — Participants in this group receive a handout called "Managing Your Mental Health" (available in Spanish and English) that provides tips on how to manage mental health through the proper maintenance of physical health and stress.
  Arms: Comparison Group

SUMMARY:
The Right Question Project-Mental Health (RQP-MH) is a three-session health education intervention that teaches clients to participate effectively in mental health care. The methodology teaches clients to identify important issues of their illness or treatment, formulate questions, and devise plans to communicate and act in effective ways that address factors impacting their mental health care, with the expectation that this behavior will increase patient-provider communication and improve the therapeutic alliance between patient and provider.

The investigators hypothesize that participants receiving the intervention will be more likely to engage and remain in mental health care, and that they will report higher activation and self-management scores as compared to control patients.

DETAILED DESCRIPTION:
The intervention is one of two Cambridge Health Alliance (CHA) projects from the University of Puerto Rico-Cambridge Health Alliance Research Center of Excellence (UPR-CHA RCE). The overall goal of the project is to evaluate an intervention that teaches patients a set of skills needed to facilitate a more active patient role in the mental health encounter, emphasizing the patient's decision-making process during mental health treatment. The project also aims to support collaborative provider-patient relationships in order to increase engagement and retention and, consequently, reduce service disparities. The intervention has been pilot-tested in the Right Question Project-Mental Health I (RQP-MH I) study (Alegría, 2008), conducted as part of the UPR-CHA EXPORT Center from September 2004 through February 2006.

The first aim of the current project is to conduct a multi-site randomized controlled trial to test the Patient Activation and Self-Management (PASM) intervention, also called RQP-MH II, in predominantly Latino mental health clinics. The investigators will assess the intervention's impact on engagement and retention in mental health care. The second aim is to explore the racial/ethnic differences in the effect of the RQP-MH II intervention for Latinos as compared to non-Latino whites, as little is known about the impact of patient race/ethnicity on the effectiveness of patient activation interventions. The fourth aim is to explore the role of patient-provider communication and therapeutic alliance as mediators of the relationship between patient activation and engagement and retention in care. It is expected that increased patient-provider communication and a stronger therapeutic alliance will result from increased participation in the decision-making process. These potential changes in the process of care are expected to consequently increase patient engagement (keeping scheduled appointments) and retention (reduction of premature unilateral termination) in mental health care.

Data shows that patients may not readily state their concerns in their medical visits (Roter et al., 1997; Korsch, Gozzi & Francis, 1968) and usually refrain from engaging in information-seeking (Beisdecker & Beisdecker, 1990). Minority patients are even less likely than their white counterparts to have a collaborative relationship with providers (Cooper-Patrick et al., 1999). This is a problematic situation particularly for minority patients, such as Latinos, who cherish maintaining a warm personal connection with their providers (American Medical Association, 1994) and may worry that bringing up questions or asking for explanations might jeopardize the relationship.

Minority patients may not be as informed about diagnosis, prognosis, and medication side effects (Schaafsma, Raynor & de Jong-van den Berg, 2003) and consequently feel disappointed that they do not receive needed information (Levinson et al., 1993). They may therefore be less compliant with treatment (Kalichman et al., 1999), and more likely to drop out of care (Takeuchi et al., 1992). Minority patients may have a less comprehensive understanding of mental health care compared to White patients (Miranda and Cooper, 2004). As a result, they are at a greater risk of assuming that the provider's decisions reflect their best interest (Flynn et al., 2004). This is exemplary of Latinos who hold traditional role expectations that oppose active involvement in the clinical encounter and prefer to delegate decisions about their care to their providers (Levinson et al., 2005; Xu, Borders & Arif, 2003).

To contend with difficulties in communication, most interventions focus on provider training (Post, Cegala & Miser, 2002), with less attention on teaching patients how to effectively express their concerns and questions to their providers (Andersen & Sharpe, 1991; Roter, 1977). Yet results from assessments of self-management of chronic conditions (Hall, Roter & Katz, 1988; Stewart et al., 1993) indicate that greater patient activation and self-management in treatment can augment satisfaction with care (Blanchard et al., 1990), improve the health care process (Rosenberg, Lussier & Beaudoin, 1997; Epstein et al., 1993), ensure the receipt of guideline concordant treatments (Clever et al., 2006), and potentially enhance health outcomes (Kaplan, Greenfield & Ware, 1989).

Most studies of patient activation and self-management in the field of mental health care have not been conducted with minority populations of low literacy nor in a language other than English. Most have not included mixed-methods (qualitative and quantitative) to evaluate the effectiveness of the intervention, and have not obtained cost information that can help evaluate whether changes in patient activation and self-management, or in treatment engagement and retention, could potentially produce savings in treatment or health care outcomes.

The proposed project is expected to fill this gap, assessing the effects of a patient activation and self-management intervention using a mixed-methods approach, with three data collection periods. The investigators hypothesize that patients participating in the patient activation and self-management intervention will be significantly more likely to engage and remain in mental health care, and will report significantly higher activation and self-management scores as compared to control patients. Given the relationship of patient participation and health outcomes, increasing Latino patient's participation in decision-making a as mechanism to eliminate service disparities is the goal of the proposed intervention.

ELIGIBILITY:
Inclusion Criteria:

* between ages of 18 and 70 (patients above age 65 will be administered the Mini-Cog, a cognitive impairment screener)
* speak English and/or Spanish
* currently receiving outpatient mental health care

Exclusion Criteria:

* suicidal ideation or attempt within the past four weeks
* lacks capacity to consent (adapted from Zayas, Cabassa, & Perez, 2005)
* only receiving services that are strictly case-management

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 724 (Actual)
Dates: Start 2008-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Patient Activation | Baseline, 30days, 90days
  Activation is defined as a behavior change approach that includes an individual's acquisition of knowledge, skills and beliefs to take thoughtful action on one's own behalf and actively participate in questions and decisions about one's health and health care treatment.
Patient Self-Management | Baseline, 30days, 90days
  Self-management focuses on patients gaining knowledge and self-efficacy to better manage their mental health condition and developing awareness of the factors that hinder or enhance their mental health outcomes.
Engagement in mental health care | Six months following last research interview
  Scheduling and keeping mental health treatment appointments over a six month period after finishing the final research interview.
Retention in mental health treatment | Six months following last research interview
  Attending four or more treatment sessions during the six month period after the final research interview (or completed treatment as designated in the medical record)

CONTACTS AND LOCATIONS:
Overall Officials: Margarita Alegria, PhD, Principal Investigator — Cambridge Health Alliance
Locations (13):
- United States (12):
  - Beth Israel Deaconness Medical Center, Boston, Massachusetts
  - Martha Eliot Health Center, Jamaica Plain, Massachusetts
  - Cambridge Health Alliance (Malden Family Medicine Center), Malden, Massachusetts
  - Cambridge Health Alliance (Central Street Health Center), Somerville, Massachusetts
  - Edward M Kennedy Health Center (Great Brook Valley Health Center), Worcester, Massachusetts
  - Community-University Health Care Center, Minneapolis, Minnesota
  - Hamm Memorial Psychiatric Clinic, Saint Paul, Minnesota
  - West Side Community Health Services - La Clinica, Saint Paul, Minnesota
  - University Behavioral Healthcare, New Brunswick, New Jersey
  - Columbia University Medical Center, Outpatient Psychiatry Program, New York, New York
  - El Futuro Clinic, Carrboro site, Carrboro, North Carolina
  - El Futuro Clinic, Durham site, Durham, North Carolina
- Clinica de Salud Mental de la Comunidad Universidad Carlos Albizu, San Juan, Puerto Rico

REFERENCES:
- [Derived] Alegria M, Carson N, Flores M, Li X, Shi P, Lessios AS, Polo A, Allen M, Fierro M, Interian A, Jimenez A, La Roche M, Lee C, Lewis-Fernandez R, Livas-Stein G, Safar L, Schuman C, Storey J, Shrout PE. Activation, self-management, engagement, and retention in behavioral health care: a randomized clinical trial of the DECIDE intervention. JAMA Psychiatry. 2014 May;71(5):557-65. doi: 10.1001/jamapsychiatry.2013.4519. PMID 24647680
- See also: Center for Multicultural Mental Health Research — http://www.multiculturalmentalhealth.org